CLINICAL TRIAL: NCT03174795
Title: A Non-Randomized, Open-Label, One Treatment, One Group Study to Investigate the Pharmacokinetics of RO7079901 and Meropenem in Patients With a Complicated Urinary Tract Infection
Brief Title: A Study to Investigate the Pharmacokinetics of RO7079901 and Meropenem in Participants With a Complicated Urinary Tract Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP39596; 2016-004478-16 (EudraCT Number)
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RO7079901 and Meropenem (Experimental): Participants will receive RO7079901 and meropenem. The duration of study drug treatment will be determined by the investigator after evaluation of the participant's response to study drug treatment. Participants should receive a minimum treatment period of 3 days and up to 14 days of intravenous (IV) study drug treatment.
  Interventions: Drug: RO7079901; Drug: Meropenem

INTERVENTIONS:
Drug: RO7079901 — Participants will receive RO7079901 2000 milligrams (mg) IV treatment, three times a day (TID) for up to 14 days.
Drug: Meropenem — Participants will receive meropenem 2000 mg IV treatment TID for up to 14 days.

SUMMARY:
This is a non-randomized, open-label, one-treatment, one group study in participants with complicated urinary tract infection (cUTI) including pyelonephritis to characterize the pharmacokinetics of RO7079901 co-administered with meropenem.

ELIGIBILITY:
Inclusion Criteria:

* Requiring hospitalization for IV antibacterial therapy for the treatment of presumed/confirmed cUTI (including pyelonephritis)
* Clinical signs and/or symptoms of pyelonephritis or a cUTI
* Urine culture taken within the 48 hours (hr) period immediately preceding the first dose of study drug contains greater than (>)1x10^5 colony forming units (CFU) per milliliter (CFU/mL) of a gram negative organism
* Negative urine pregnancy test result confirmed by a blood test
* Agreement to remain abstinent or use a contraceptive method

Exclusion Criteria:

* Has a concomitant infection requiring antibacterial therapy, in addition to study drug
* Confirmed fungal urinary tract infection
* Moderate or severe renal impairment, or end-stage renal disease requiring renal replacement therapy or a recipient of a renal transplant
* Documented presence of immunodeficiency, or a severely immunocompromised condition or use of systemic immunosuppressant therapy
* Any rapidly progressing disease or immediately life-threatening illness, or other terminal illness or condition with high risk of mortality meaning that the participant is considered, in the opinion of the Investigator, unlikely to survive the study period
* Urinary tract surgery or clinically significant urogenital trauma in the one week immediately preceding study entry
* Urinary tract infection (UTI) symptoms potentially attributable to another process (sexually transmitted infections or prostatitis)
* Suspected or confirmed perinephric or intra renal abscess
* Complete obstruction of any portion of the urinary tract, or a permanent urinary diversion
* History of epilepsy, brain lesions or other significant neurological disorders
* Use of probenecid within the 7 days before enrollment
* Known history of clinically significant hypersensitivity or severe allergic reaction to meropenem or any other antibiotic
* Any other ongoing condition or disease, or clinically significant abnormalities in laboratory test results that the investigator considers would render the participant unsuitable for the study
* Women who are pregnant, planning to become pregnant, or lactating
* Participation in a clinical study of an investigational drug or device within one month prior to enrollment
* Prior enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-16 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve Over the Dosing Interval (AUC0-tau) of RO7079901 | Pre-dose (0 hr), 1.5 hr (end of infusion [infusion duration=1.5 hr]), 3, 4.5, 6, 8 hr post dose on Days 1, 3; pre-dose (0 hr), 1.5 and 8 hr post dose on Days 5 and 7
Total Clearance (CL) of RO7079901 | Pre-dose (0 hr), 1.5 hr (end of infusion [infusion duration=1.5 hr]), 3, 4.5, 6, 8 hr post dose on Days 1, 3; pre-dose (0 hr), 1.5 and 8 hr post dose on Days 5 and 7
Renal Clearance (CLr) of RO7079901 | Days 1 and 3 (all urine passed in the 8-hour period after morning dose will be collected)
Maximum Observed Plasma Concentration (Cmax) of RO7079901 | Pre-dose (0 hr), 1.5 hr (end of infusion [infusion duration=1.5 hr]), 3, 4.5, 6, 8 hr post dose on Days 1, 3; pre-dose (0 hr), 1.5 and 8 hr post dose on Days 5 and 7
Cumulative Amount Excreted in Urine Over the Dosing Interval (Ae) of RO7079901 | Days 1 and 3 (all urine passed in the 8-hour period after morning dose will be collected)
Fraction Excreted into the Urine (Fe) of RO7079901 | Days 1 and 3 (all urine passed in the 8-hour period after morning dose will be collected)
Time of Maximum Observed Plasma Concentration (Tmax) of RO7079901 | Pre-dose (0 hr), 1.5 hr (end of infusion [infusion duration=1.5 hr]), 3, 4.5, 6, 8 hr post dose on Days 1, 3; pre-dose (0 hr), 1.5 and 8 hr post dose on Days 5 and 7
Steady State Volume of Distribution (Vss) of RO7079901 | Pre-dose (0 hr), 1.5 hr (end of infusion [infusion duration=1.5 hr]), 3, 4.5, 6, 8 hr post dose on Days 1, 3; pre-dose (0 hr), 1.5 and 8 hr post dose on Days 5 and 7

SECONDARY OUTCOMES:
AUC0-tau of Meropenem | Pre-dose (0 hr), 1.5 hr (end of infusion [infusion duration=1.5 hr]), 3, 4.5, 6, 8 hr post dose on Days 1, 3; pre-dose (0 hr), 1.5 and 8 hr post dose on Days 5 and 7
CL of Meropenem | Pre-dose (0 hr), 1.5 hr (end of infusion [infusion duration=1.5 hr]), 3, 4.5, 6, 8 hr post dose on Days 1, 3; pre-dose (0 hr), 1.5 and 8 hr post dose on Days 5 and 7
CLr of Meropenem | Days 1 and 3 (all urine passed in the 8-hour period after morning dose will be collected)
Cmax of Meropenem | Pre-dose (0 hr), 1.5 hr (end of infusion [infusion duration=1.5 hr]), 3, 4.5, 6, 8 hr post dose on Days 1, 3; pre-dose (0 hr), 1.5 and 8 hr post dose on Days 5 and 7
Ae of Meropenem | Days 1 and 3 (all urine passed in the 8-hour period after morning dose will be collected)
Fe of Meropenem | Days 1 and 3 (all urine passed in the 8-hour period after morning dose will be collected)
Tmax of Meropenem | Pre-dose (0 hr), 1.5 hr (end of infusion [infusion duration=1.5 hr]), 3, 4.5, 6, 8 hr post dose on Days 1, 3; pre-dose (0 hr), 1.5 and 8 hr post dose on Days 5 and 7
Vss of Meropenem | Pre-dose (0 hr), 1.5 hr (end of infusion [infusion duration=1.5 hr]), 3, 4.5, 6, 8 hr post dose on Days 1, 3; pre-dose (0 hr), 1.5 and 8 hr post dose on Days 5 and 7

CONTACTS AND LOCATIONS:
Locations (14):
- United States (2):
  - eStudySite, La Mesa, California
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
- Hungary (3):
  - Semmelweis University, First Dept of Medicine, Budapest
  - Szent Imre Egyetemi Oktatokorhaz, Budapest
  - Kenezy Gyula Korhaz-Rend. Eges. Szol.; Klinikai Farm. Infek. es Allerg. Intezet, Debrecen
- Latvia (3):
  - Liepaja Regional hospital, Liepāja
  - P.Stradina Kliniska Uni Tes Slimnica; Latvian Center of Nephrology, Riga
  - Riga East clinical university hospital, Riga
- Poland (3):
  - Klinika Urologii Ogólnej: Collegium Medicum Uniwersytetu Mikołaja Kopernika w Toruniu; Urology, Bydgoszcz
  - Uniwersytecki Szpital Kliniczny im WAM CSW; Klinika Nefrologii i Transplantologii Nerek, Lodz
  - Szpital Kliniczny Dzieciątka Jezus; Oddział Urologii, Warsaw
- Serbia (3):
  - Clinical Center of Serbia; Clinic of Urology, Belgrade
  - Clinical Center Zemun, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade